CLINICAL TRIAL: NCT06352385
Title: A Comprehensive Epidemiological Investigation of Malocclusion in China
Brief Title: Epidemiological Investigation of Malocclusion in China
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Bing Fang, Professor, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SH9H-2024-TK16-1.0
Record Dates: First submitted 2024-03-22; First posted 2024-04-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Epidemiological Investigation; Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Children aged 4 -6: This is a non intervention-observation only study.
- Children aged 9 -11: This is a non intervention-observation only study.
- Students aged 13 -15: This is a non intervention-observation only study.
- Students aged 17-20: This is a non intervention-observation only study.

SUMMARY:
Malocclusion is a kind of craniomaxillofacial complex deformity caused by heredity, environment, bad habits, trauma, inflammation, tumor and aging. Notably, the last comprehensive national prevalence data on malocclusion in China, which encompassed a significant sample size, dates back over two decades. Given the evolving nature of these epidemiological metrics, such as prevalence rates, it is imperative to update our understanding. Consequently, there is an urgent need for China to undertake a unified, standardized epidemiological survey of malocclusion with a substantial sample size to ensure accurate and timely data collection.

DETAILED DESCRIPTION:
With the improvement of our country's living and cultural level, orthodontic treatment for malocclusion has emerged as a critical need that significantly impacts individuals' physical and mental wellbeing, as well as their social life in contemporary society. To obtain the prevalence rate, demand index and risk factor analysis of malocclusion in China serves as a fundamental prerequisite for effective diagnosis, identifying the optimal treatment window, and devising tailored treatment plans.

The purpose of this study is as follows:

1. Obtaining epidemiological data such as the prevalence rate of malocclusion is the cornerstone of prevention and treatment of malocclusion, and is also the prerequisite of carrying out a series of studies;
2. Establishing China's orthodontic treatment demand index offers vital support for the advancement of orthodontics and oral healthcare.;
3. Updating and enhancing X-ray head image measurement normal reference value provides a more scientific and objective foundation for orthodontic planning, improves the level of diagnosis and treatment, and fosters the development of related disciplines.

The implementation of this project will not only foster an improvement in the overall oral health of the populace but also establish a scientific foundation for oral medicine research and the development of prevention and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with all genders;
2. Individuals with good general health;
3. Individuals with no history of orthodontic treatment or other maxillofacial surgical interventions;
4. Individuals who agree to and are willing to sign the informed consent form.

Exclusion Criteria:

1. Individuals diagnosed with genetic or systemic disorders;
2. Individuals with a recent (within the past 3 months) history of maxillofacial trauma;
3. Individuals who are incapable of undergoing oral examinations or completing the necessary questionnaires.

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study included four age groups: students aged 4-6 years (senior grade of kindergarten),9-11 years (fourth grade in primary school),13-15 years (eighth grade),and 17-20 years (freshman in college).
Sampling Method: Probability Sample
Enrollment: 19847 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The Prevalence rate of malocclusion | recruitment until December 2026
  The Index of Orthodontic Treatment Need and Dental Aesthetic Index were used to record the Malocclusion deformities,The Index of Orthodontic Treatment Need or Dental Aesthetic Index ≥3 is recorded as Malocclusion.The prevalence rate of malocclusion was the number of cases of Malocclusion /the total number of investigated cases during the research investigation.

SECONDARY OUTCOMES:
Dental Aesthetic Index of each age group | recruitment until December 2026
  Fill in the questionnaire through clinical examination,then calculate Dental Aesthetic Index according to the results of the questionnaire
Index of Orthodontic Treatment Need of each age group | recruitment until December 2026
  Fill in the questionnaire through clinical examination,then calculate Index of Orthodontic Treatment Need according to the results of the questionnaire

OTHER OUTCOMES:
dietary habit | recruitment until December 2026
  Questionnaire survey
oral hygiene habits | recruitment until December 2026
  Questionnaire survey
Bad oral habit | recruitment until December 2026
  Questionnaire survey

CONTACTS AND LOCATIONS:
Overall Officials: Bing Fang, PhD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University

IPD SHARING:
Plan to Share IPD: No